CLINICAL TRIAL: NCT05460533
Title: Phase II Open Label Multicenter Study of Early REinFusion of Tisagenlecleucel to Promote DUrable B-CEll ApLasia in Pediatric and Young Adult Patients With Relapsed/Refractory CD19-Positive B-Cell Acute Lymphoblastic Leukemia (REFUEL)
Brief Title: A Second Infusion (Early Reinfusion) of Tisagenlecleucel in Children and Young Adults With B-Cell Acute Lymphoblastic Leukemia(B-ALL)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-220
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: Tisagenlecleucel; Relapsed/Refractory CD19-Positive B-Cell; REinFusion; REFUEL; 22-220
MeSH Terms: conditions — Burkitt Lymphoma; Recurrence | interventions — tisagenlecleucel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tisagenlecleucel (Experimental): Patients will receive reinfusion of tisagenlecleucel on day +30-60 after their initial infusion if meeting eligibility criteria. Tisagenlecleucel is an autologous cellular immunotherapy product that is comprised of CD3+T cells that have undergone ex vivo T cell activation, gene modification, expansion, and formulation in infusible cryomedia.
  Interventions: Biological: Tisagenlecleucel

INTERVENTIONS:
Biological: Tisagenlecleucel — Tisagenlecleucel will be infused based on institutional guidelines. Reinfusion of tisagenlecleucel will occur 30-60 days following the first dose.

SUMMARY:
The researchers are doing this study to see if early reinfusion of tisagenlecleucel can keep participants in B-CEll ApLasia at 6 months after their first infusion. The researchers will also look at the safety of early reinfusion and how effective it is at treating B-ALL.

DETAILED DESCRIPTION:
Prior to initial tisagenlecleucel cell infusion, lymphodepleting chemotherapy (LDC) is required with standard dosing cyclophosphamide and fludarabine as per standard-of-care (fludarabine 30mg/m^2 /dose x 4 doses and cyclophosphamide 500mg/m^2 /dose x 2 doses). Dose adjustments based off ideal body weight (IBW) and/or per institutional guidelines are allowed. LDC should be completed 2 to 14 days prior to the first tisagenlecleucel infusion. LDC may be repeated in cases where tisagenlecleucel has been delayed by more than 4 weeks. No additional LDC will be given prior to the early reinfusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with R/R B-ALL who have received commercial tisagenlecleucel and have (an) additional dose(s) available for early reinfusion
* History of CD19 expressing (in peripheral blood or bone marrow by flow cytometry) BALL prior to tisagenlecleucel infusion
* Peripheral blood B-cell aplasia (BCA) within 14 days prior to reinfusion (See section 13.8: B-cell aplasia will be defined as peripheral blood (PB) absolute B lymphocyte count ≤ 50/μL. If BCA evaluation is repeated at any timepoint prior to reinfusion, it must be negative to proceed with reinfusion
* Minimal residual disease negative complete remission (CR/CRi) in bone marrow within 14 days prior to reinfusion, including resolution of extramedullary disease
* Patients with tisagenlecleucel that is deemed out of specification (OOS) will be permitted on this protocol if the reason for OOS is deemed to not impact the toxicity and efficacy profile of CAR T cell therapy

  °Reasons for product being OOS include cell viability < 80%, total nucleated cell count <2 × 10^9 in leukapheresis product, failed interferon-γ release assay, leukapheresis product collected >9 months prior, and determination of residual beads >50 beads per 3 × 10^6 cells
* Patients age: < 26 years at time of first tisagenlecleucel order placement
* Recovered from severe toxicities following initial dose of tisagenlecleucel

  * CRS
  * Neurotoxicity/ICANS
* Adequate organ function at time of treatment is required and is defined:

  * Hepatic: Serum bilirubin ≤ 2 mg/dL, unless benign congenital hyperbilirubinemia
  * Hepatic: AST and ALT < 5x the upper limit of normal for age, unless thought to be disease-related
  * Renal: Serum creatinine <1.5x normal for age. If serum creatinine is outside the normal range, then CrCl > 60 mL/min/1.73m2 (calculated or estimated) or GFR (mL/min/1.72m2 ) >55% of predicted normal for age

Age Mean GFR +/-SD (mL/min/1.73 m2)

* 1 week 40.6 + / - 14.8
* 2 - 8 weeks 65.8 + / - 24.8
* > 8 weeks 95.7 +/- 21.7
* 2 - 12 years 133 +/- 27
* 13 - 21 years (males) 140 +/- 30
* 13 - 21 years (females) 126.0 + / - 22.0 Abbreviations: GFR, glomerular filtration rate; SD, standard deviation. Greater than 2 years old: Normal GFR is 100 mL/ min. Infants: GFR must be corrected for body surface area.

  * Cardiac: LVEF ≥ 50% by multi-gated acquisition scan (MUGA), resting echocardiogram, or cardiac magnetic resonance imaging (MRI) within 6 weeks of screening
  * Pulmonary: Oxygen saturation as recorded by pulse oximetry of ≥ 90% on room air
* Adequate performance status:

  * Age ≥ 16 years: ECOG ≤ 1 or Karnofsky > 60% at treatment
  * Age < 16 years: Lansky > 60% at treatment
* Patient must be enrolled on institutional CIBMTR reporting protocol for immune effector cells (IEC)/CAR T cells
* Each patient must be willing to participate as a research subject, and patient or legal guardian must sign an informed consent form, along with patient assent if between 7 to 17 years of age. Legally authorized representatives of adult patients with impaired decision-making capacity will also be able to sign consent.

Exclusion Criteria:

* Greater than 60 days from first tisagenlecleucel infusion
* Ongoing severe toxicities from initial CAR T cell infusion
* Received non-standard lymphodepleting chemotherapy (LDC) prior to initial tisagenlecleucel dose
* Standard LDC is defined as:

  * Fludarabine 30mg/m^2/dose x 4 doses
  * Cyclophosphamide 500mg/m^2/dose x 2 doses
* Loss of BCA at any timepoint prior to reinfusion
* Clinically significant active infection confirmed by clinical evidence, imaging, or positive laboratory tests (e.g., blood cultures, PCR for DNA/RNA, etc.)
* Patient/parent/guardian unable to give informed consent or unable to comply with the treatment protocol
* Pregnant or lactating women; women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception while taking study treatment and for at least 12 months after the tisagenlecleucel infusion and until CAR T-cells are no longer present by flow cytometry on two consecutive tests.
* Sexually active males, unless they are willing to use a condom during intercourse while taking study treatment and for at least 12 months after the tisagenlecleucel infusion and until CAR T-cells are no longer present by flow cytometry on two consecutive tests.
* Other uncontrolled, symptomatic, intercurrent illness including but not limited to infection, psychiatric illness, or social situations that would limit compliance with study requirements or in the opinion of the PI would pose an unacceptable risk to the subject
* Any other issue which, in the opinion of the treating physician, would make the patient ineligible for the study

Ages: 1 Day to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
decrease the loss of peripheral BCA rate | 6 months
  below 10% (from 26% to 9%)

SECONDARY OUTCOMES:
number and percentage of toxicities with early reinfusion of CAR T cells | 1 year
  CTCAE Version 5 will be utilized for toxicity evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Curran, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Children's Hospital of Los Angeles (Data Collection Only), Los Angeles, California
  - Stanford University (Data Collection Only), Stanford, California
  - Children's Hospital Colorado (Data Collection Only), Aurora, Colorado
  - Johns Hopkins University (Data Collection Only), Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center (Data Collection Only), Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm